CLINICAL TRIAL: NCT00423007
Title: Efficacy and Safety of Topical Bromfenac Ophthalmic Solution vs. Placebo in Subjects With a History of Allergic Conjunctivitis
Brief Title: Efficacy and Safety of Topical Bromfenac Ophthalmic Solution vs. Placebo in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTA-BR-CS03
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bromfenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromfenac (Experimental): Ophthalmic Solution
  Interventions: Drug: Bromfenac
- Placebo (Placebo Comparator): Vehicle ophthalmic solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bromfenac
  Arms: Bromfenac
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the efficacy and safety of bromfenac ophthalmic solution for treatment in subjects with a history of allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* History of clinically active allergic conjunctivitis
* Agree to return for all required visits
* Agree to avoid disallowed meds

Exclusion Criteria:

* Known hypersensitivity to bromfenac and salicylates

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Treatment of ocular itching

SECONDARY OUTCOMES:
Treatment of chemosis, episcleral and ciliary hyperemia, ocular mucous discharge, eyelid swelling, foreign body sensation, nasal symptoms, and/or tearing

CONTACTS AND LOCATIONS:
Overall Officials: Jon Williams, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States